CLINICAL TRIAL: NCT02752724
Title: Ketamine vs. Methohexital Anesthesia for Improvement of Major Depressive Disorder in Electroconvulsive Therapy
Brief Title: Ketamine Anesthesia for Improvement of Depression in ECT
Acronym: KAID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. Charles William Carspecken, MD, MBA, MSc, Physician --Anesthesiologist, VA Puget Sound Health Care System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00850
Record Dates: First submitted 2016-03-25; First posted 2016-04-27 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Major Depressive Disorder
Keywords: major depressive disorder; electroconvulsive therapy; metabolomics; treatment resistant depression; anesthesiology; ketamine; prospective randomized clinical trial
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant | interventions — Ketamine; Methohexital

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine Interventional Arm (Experimental): 1.0 mg/kg IV ketamine (experimental arm) intravenously (IV) for the duration of their ECT index course over 2-3 weeks
  Interventions: Drug: Ketamine
- Methohexital Control Arm (Active Comparator): 1mg/kg of methohexital (standard arm) intravenously (IV) for the duration of their ECT index course over 2-3 weeks
  Interventions: Drug: Methohexital

INTERVENTIONS:
Drug: Ketamine — Ketamine anesthesia for ECT index course with measurement cerebral metabolic regional oximetry, EEG seizure quality, cognitive scoring and serum metabolites.
  Other Names: Ketalar
  Arms: Ketamine Interventional Arm
Drug: Methohexital — Methohexital anesthesia for ECT index course with measurement cerebral metabolic regional oximetry, EEG seizure quality, cognitive scoring and serum metabolites.
  Other Names: Brevital
  Arms: Methohexital Control Arm

SUMMARY:
The purpose of this prospective randomized clinical trial is to determine if patients receiving ketamine as a part of general anesthesia during electroconvulsive therapy (ECT) rather than standard of care will have improvement in symptoms of depression after a course of ECT treatments. The investigators hypothesize that utilization of ketamine for induction of general anesthesia during ECT treatments will improve symptoms of depression better than standard care.

This study is ONLY open to patients eligible to receive healthcare services through the Department of Veterans Affairs at the VA Puget Sound, which means service in the active military, naval or air service or separation under any condition other than dishonorable. Qualifications for VA health care benefits can be found at va.gov.

DETAILED DESCRIPTION:
The purpose of this prospective randomized clinical trial is to determine if patients receiving ketamine as a part of general anesthesia during electroconvulsive therapy (ECT) rather than standard of care will have improvement in symptoms of depression after a course of ECT treatments. The investigators hypothesize that utilization of ketamine for induction of general anesthesia during ECT treatments will improve symptoms of depression better than standard care.

For induction of general anesthesia for ECT, patients will receive either 1mg/kg of methohexital (standard arm) or 1.0 mg/kg IV ketamine (experimental arm) intravenously (IV) for the duration of their ECT index course over 2-3 weeks. The primary outcome in this trial is change in symptoms of depression assessed by standard questionnaires: Patient Health Questionnaire 9 (PHQ9) and Hamilton Depression Rating Scale (HAM-D) score changes from baseline and final ECT administration. Secondary outcomes are changes in cognitive status as assessed by the Montreal Cognitive Assessment (MoCA) scale, quality of seizures and after seizure, changes in serum metabolites (including kynurenine, D/L-serine and other glutamate intermediates) after treatment and need for further ECT courses (relapse) within 1 year after initial course.

Approximately 50 veterans with the diagnosis of major depressive disorder older than 18 years of age undergoing ECT will be randomized and blinded to the intervention. Operative ECT clinicians will not be blinded; clinicians evaluating patients will be blinded. Exclusion criteria for this study include uncontrolled hypertension, blood pressure > 180/90 mmHg at the pre-anesthesia clinic visit, renal failure, neurologic disorders (e.g. epilepsy, space occupying lesions, traumatic brain injuries in the past 6 months), myocardial infarction in the past 6 months, known allergies or adverse reactions to ketamine, American Society of Anesthesiology Physical Class greater than 3, concomitant psychosis, schizophrenia or current abuse of alcohol or illicit substances and pregnancy.

The long term objective of this trial is to systematically characterize ketamine's effect on depression outcomes utilizing validated scoring tools, its safety profile throughout an ECT index course, ketamine's effect on seizure quality and changes in novel translational endpoints to better understand mechanisms of action of ketamine and its potential role in treatment of psychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

* outpatients or inpatients at the Puget Sound VA with diagnosis of major depressive disorder or bipolar 1 or 2 over the age of 18 undergoing index course ECT

Exclusion Criteria:

* uncontrolled hypertension (blood pressure > 180/90 mmHg at the pre-anesthesia clinic visit)
* renal failure
* neurologic disorders (e.g. epilepsy, space occupying lesions, traumatic brain injuries in the past 6 months)
* myocardial infarction in the past 6 months
* known allergies or adverse reactions to ketamine
* American Society of Anesthesiology Physical Class greater than 3
* concomitant psychosis
* schizophrenia or current abuse of alcohol or illicit substances and pregnancy (any trimester)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Depression Patient Health Questionnaire 9 (PHQ9) Scoring | Change from Baseline Score 24 hours prior to starting ECT to PHQ9 score 72 hours following last ECT session
  Evaluate the efficacy and safety of repeat anesthetic ketamine dosing during a complete index course of ECT compared with methohexital using change in a validated depression scoring tool (Patient Health Questionnaire 9) administered 24 hours prior to starting an ECT index course treatment (baseline) with a PHQ9 score 72 hours after the last/final ECT session for approximately fifty patients. The PHQ9 Scoring ranges from 0 to 27 in order to monitor depression severity over time for newly diagnosed patients or patients in current treatment for depression.

SECONDARY OUTCOMES:
Soluble Amino Acid Metabolomic Biomarkers | 30 minutes prior to first ECT session and within 30 minutes after final ECT session
  Measurement of biomarkers before/after ECT index course serum aqueous metabolites from patient venous blood drawn from intravenous line specifically concentration of serine, tryptophan, quinolinic acid, kynurenine in mcg/dL using mass spectrometry. Samples are collected 30 minutes prior to first ECT session and within 30 minutes after final ECT treatment session.
ECT Seizure Duration | Length of each intraoperative ECT seizure during an index course typically 6-12 individual seizures measure from start of seizure in operating room to end of seizure in operating room.
  This trial will measure intra-operative seizure length/duration (in seconds) using a standard ECT machine which helps the ECT machine operator determine the total length of time a patient is seizing during each ECT seizure session. An index course of ECT treatment typically involves 6 to 12 seizures titrated to a patient's response. The investigators will record the length of seizure for every treatment session for every patient.
Change in Montreal Cognitive Assessment (MoCA) Scoring | Change from Baseline Score 24 hours prior to starting ECT to MoCA score 72 hours following last ECT session
  Evaluate the efficacy and safety of repeat anesthetic ketamine dosing during a complete index course of ECT compared with methohexital using change in a validated cognitive scoring tool (Montreal Cognitive Assessment MoCA) administered 24 hours prior to starting an ECT index course treatment (baseline) with a MoCA score 72 hours after the last/final ECT session for approximately fifty patients. The MoCA Scoring ranges from 0 to 30 in order to rapidly screen for mild cognitive dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Borisovskaya, MD, Study Director — Puget Sound VA Medical Center, Dept of Psychiatry; Irene Rozet, MD, Principal Investigator — Puget Sound VA Medical Center, Dept of Anesthesiology
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No